CLINICAL TRIAL: NCT03239301
Title: Robotic-assisted Upper Extremity Training in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Timur Ekiz, Medical Doctor, Physical and Rehabilitation Medicine Specialist, Ankara Physical Medicine and Rehabilitation Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1240
Record Dates: First submitted 2017-07-31; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Spinal Cord Injury Cervical

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Rehabilitation (Active Comparator): Conventional rehabilitation program consisted range of motion (ROM) exercises, balance and coordination training, progressive resistive exercises, posture training, gait training, and occupational therapy as much as the patients tolerated. Conventional rehabilitation was tailored to the patient considering his requires and expectancies.
  Interventions: Procedure: Conventional Rehabilitation
- Robotic Rehabilitation + Conventional Rehab (Active Comparator): The Armeo Spring HocomAG Inc. (Volketswil, Switzerland) device was used in robot assisted upper limb rehabilitation program. A
  Interventions: Procedure: Conventional Rehabilitation; Procedure: Robotic REhabilitation

INTERVENTIONS:
Procedure: Conventional Rehabilitation — Conventional rehabilitation program consisted range of motion (ROM) exercises, balance and coordination training, progressive resistive exercises, posture training, gait training, and occupational therapy as much as the patients tolerated. Conventional rehabilitation was tailored to the patient considering his requires and expectancies.
Procedure: Robotic REhabilitation — The Armeo Spring HocomAG Inc. (Volketswil, Switzerland) device was used in robot assisted upper limb rehabilitation program. Assistive component of the robotic arm was adjusted in accordance with motor level of each patient. Variety and difficulty of games were chosen according to the ability and functional status of the patients. Variety and difficulty level of the games were modified according to progress of patients by the same physiotherapist.
  Arms: Robotic Rehabilitation + Conventional Rehab

SUMMARY:
Study design: Controlled Trial Objective: To evaluate the effectiveness of robotic-assisted training of forearm and hand functions in spinal cord injury patients Setting: Ankara Physical Medicine and Rehabilitation Training and Research Hospital, Turkey Methods: Forty patients were allocated into robotic and control groups. Both groups received conventional rehabilitation program for four weeks. Moreover, robotic group received robotic rehabilitation program tailored to the patient five times a week (each session of 30 min).

Baseline data and post-intervention data was compared.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 18-50
* Cervical Level of Spinal Cord Injury

Exclusion Criteria:

* Severe upper extremity contractures in the joints
* Intensive spasticity (Ashworth 3-4)
* Shoulder pain that causes exercise intolerance

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | Four weeks
  Scale Evaluating the Functionality
Spinal Cord Independence Measure III | Four weeks
  Scale Evaluating the Functionality and independence
Short Form-36 | Four weeks
  Scale Evaluation the activities of daily living

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Fizik Tedavi ve REhabilitasyon Eğitim ve Araştırma Hastanesi, Ankara
  - Ankara Physical MEdicine and REhabilitation Trainign and Research Hospital, Ankara

IPD SHARING:
Plan to Share IPD: Undecided